CLINICAL TRIAL: NCT06686017
Title: A Prospective Post-Market Historically Controlled Open-Label Study to Assess the Efficacy of Virtuos in Lumbar Fusion
Brief Title: Virtuos Bone Graft in Lumbar Fusion
Status: Enrolling by invitation | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-VBG-24
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease
Keywords: Lumbar spinal fusion; Cellular based allograft; Anterior lumbar interbody fusion (ALIF); Lateral lumbar interbody fusion (LLIF); Virtuos
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with one or two level degenerative disc disease of the lumbar spine: There are no investigational interventions. Subjects will undergo a one or two level spinal fusion procedure per the attending physician/surgeon standard practice.

SUMMARY:
A post-market open label study to assess the efficacy of a cellular based allograft bone graft in lumbar spinal fusion at one or two levels

DETAILED DESCRIPTION:
Single arm prospectively enrolled observational study of subjects who undergo lumbar spinal fusion at one or two levels with an anterior or lateral surgical approach using a cellular based allograft (Virtuos) as the bone graft There is no experimental intervention for this study. Subjects will be treated per standard of care by their attending physician/surgeon. The primary endpoint in this study is fusion success at 12 months. as determined by the attending physician/surgeon using CT as the imaging modality. The fusion rates observed at 12-months will be compared to an historical group of patients that underwent a one or two level lumbar fusion procedure with an anterior or lateral approach using a cellular based allograft (Trinity Elite).

ELIGIBILITY:
Inclusion Criteria:

Subject must be 18 years of age (≥ 18 years) or older at the time of consent.

* Subject must undergo lumbar interbody fusion study at 1-2 contiguous levels.
* Virtuos must be the primary bone graft (≥ 50% of the total graft volume) and may be augmented with autograft or cortical or cancellous bone chips.
* Subject must be willing and able to sign an informed consent document.
* Subject must be willing and able to return for all follow-up visits, agree to participate in postoperative clinical and radiographic evaluations, and comply with the required study protocol.-

Exclusion Criteria:

* Subject is under 18 years of age (<18) at the time of consent.

  * Subject has had prior lumbar spine fusion surgery at any level.
  * Subject has greater than grade 1 spondylolisthesis of the lumbar spine. Subject is currently undergoing treatment for malignancy or has undergone treatment for malignancy in the past 5 years (benign skin cancer is permitted)
  * Subject has an active local or systemic infection or is undergoing adjunctive treatment for local or systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are patients with degenerative disc disease of the lumbar spine at one or two levels who are considered to be candidates for spinal fusion surgery by their attending physician/surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Fusion | 12-months
  Fusion of the spinal motion segments

SECONDARY OUTCOMES:
Disability (ODI) | 12 months
  The ODI will be used to assess disability if the patient reported outcomes are routinely collected at participating centers.
Pain (NPRS) | 12 months
  A pain rating scale (VAS or NRS) will be used to assess pain levels at baseline and follow-up visits, if pain assessment is routinely collected as standard of care at participating sites. 0 will indicate no pain and 10 will indicate the highest amount of pain possible.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - South Bend Orthopaedics, South Bend, Indiana
  - Michigan Orthopedic Surgeons, Southfield, Michigan
  - Northern Rockies Orthopaedics, Missoula, Montana
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - OrthoSC, Myrtle Beach, South Carolina
  - Lowcountry Orthopaedics and Sports Medicine, North Charleston, South Carolina
  - South Carolina Sports Medicine, North Charleston, South Carolina
  - UT Southwestern Medical Center, Frisco, Texas
  - Tuckahoe Orthopaedics, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided